CLINICAL TRIAL: NCT00335478
Title: Phase II Open Label Pilot Trial of Empiric Daptomycin Treatment for Oncology Patients With Neutropenic Fever
Brief Title: Daptomycin in Treating Neutropenia and Fever in Patients With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000476568; OHSU-CPC-05052-L (Other: OHSU Knight Cancer Institute); OHSU-1321 (Other: OHSU IRB); CUBIST-OHSU-CPC-05052-L (Other: Cubist Pharmaceuticals)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Fever; Sweating; Hot Flashes; Infection; Neutropenia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neutropenia; infection; unspecified adult solid tumor, protocol specific; fever, sweats, and hot flashes
MeSH Terms: conditions — Fever; Hot Flashes; Infections; Neutropenia | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daptomycin (Experimental)
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — daptomycin 6 mg/kg over 30 minutes every 24 hours until patient is afebrile and ANC is >500 cells/mm^3.
  Other Names: Cubicin

SUMMARY:
RATIONALE: Antibiotics, such as daptomycin, may control neutropenia, fever, and infection in patients with cancer.

PURPOSE: This phase II trial is studying how well daptomycin works in treating neutropenia and fever in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the response rate to therapy within 72 hours of starting daptomycin in cancer patients with neutropenic fever.

Secondary

* Assess the percentage of bacterial cures in patients with documented gram-positive bacterial infections.
* Assess time to afebrile state.
* Assess the pharmacokinetic data of daptomycin in neutropenic patients.
* Document the incidence of breakthrough infections that require a change of therapy or additional agents to clear.
* Assess the tolerability of daptomycin in neutropenic patients.
* Assess and document adverse events and toxicity due to daptomycin.

OUTLINE: This is an open-label, pilot study.

Patients first receive standard treatment for gram-negative bacteria for 72 hours. If the patient is still febrile at 72 hours, daptomycin is administered.

Patients receive daptomycin IV over 30 minutes once daily. Patients who are afebrile, not neutropenic (absolute neutrophil count [ANC] > 500/mm³), and have no signs of infection after 72 hours of therapy may discontinue daptomycin. Patients who are afebrile and neutropenic (ANC < 500/mm³) after 72 hours of therapy continue to receive daptomycin until absolute neutrophil count (ANC) > 500/mm³ for 2 consecutive days. Patients who are febrile with or without continued neutropenia (ANC < 500/mm³) after 72 hours of therapy continue to receive daptomycin for up to 10-14 days in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Diagnosis of neutropenic fever

  * Temperature > 38.3°C once OR ≥ 38°C twice within 12 hours
  * Absolute neutrophil count < 500/mm^³ and ≥ 1 of the following:

    * Mucositis
    * Concurrent skin or soft tissue infection
    * Indwelling catheter and/or suspected catheter infection
    * Recent quinolone prophylaxis
    * Positive blood cultures for gram-positive cocci before final identification or other documented gram-positive pathogen
    * Colonization with β-lactam resistant gram-positive organisms (commonly the nares or the skin)
    * Hypotension, tachycardia, narrowed pulse pressures, tachypnea, or other signs of cardiovascular compromise
  * Expected duration of neutropenia ≥ 3 days
* No known infection with daptomycin-resistant organism or gram-negative organism and not yet meeting criteria for the addition of gram-positive antimicrobial therapy
* No suspected meningitis or osteomyelitis
* No documented or suspected gram-positive pneumonia
* No suspected or proven endocarditis

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 2 weeks
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception
* No known sensitivity to daptomycin or product excipients
* No history of or concurrent rhabdomyolysis
* No HIV positivity
* No psychiatric disorders that would preclude study compliance
* No signs or symptoms of myopathy with creatine phosphokinase (CPK) elevation > 1,000 U/L (5 times upper limit of normal [ULN])

  * No CPK elevations > 10 times ULN in patients with no signs or symptoms of myopathy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 7 days since prior daptomycin or other antibiotic agents covering gram-positive organisms
* No concurrent hemodialysis or continuous ambulatory peritoneal dialysis
* No concurrent succinylcholine, ethanol, fludrocortisone, olanzapine, or pioglitazone
* No concurrent hydroxymethyl glutaryl (HMG) coenzyme A (HMG CoA) reductase inhibitors (e.g., lovastatin, simvastatin, atorvastatin)
* Concurrent therapy for gram-negative bacterial infection allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin: 6 mg/kg over 30 minutes every 24 hours until patient is afebrile and ANC is >500 cells/mm^3.
Period: Overall Study
Arm/Group | Daptomycin
Started | 54
Completed | 30
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Daptomycin
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age, Continuous [Median (Standard Deviation); unit: years] | 50.4 (16.730)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Became Afebrile Within 72 Hours of Starting Daptomycin.
Description: If after 72 hours of daptomycin treatment, the patient is afebrile and has absolute neutrophil count (ANC) >500 cells/mm^3 for 48 hours with no site of infection, negative cultures, and no clinical indications for therapy, the antibiotic regimen will be discontinued.
  Complete Response: Resolution of fever and clinical signs/symptoms of infection.
  Partial Response: Resolution of fever without resolution of clinical signs of infection.
Time Frame: Within 72 hours of starting daptomycin
Measure: Number; unit: participants
Arm/Group | Daptomycin
Number analyzed (Participants) | 30
participants | 16

ADVERSE EVENTS:
Arm/Group | Daptomycin
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No